CLINICAL TRIAL: NCT01055223
Title: The Association Between Exposure to Spironolactone or Amiloride and Fracture Risk Among Subjects Treated With Thiazolidinediones
Brief Title: Fracture Risk With Thiazolidinediones
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113332
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Fractures, Bone; Type II Diabetes
Keywords: thiazolidinediones; rosiglitazone; amiloride; pioglitazone; fracture; Spironolactone
MeSH Terms: conditions — Fractures, Bone; Diabetes Mellitus, Type 2 | interventions — Pemoline; Troglitazone; Spironolactone; Amiloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes subjects: Type 2 diabetes subjects
  Interventions: Drug: TZD only (RSG or PIO or troglitazone); Drug: TZD + spironolactone; Drug: TZD + amiloride

INTERVENTIONS:
Drug: TZD only (RSG or PIO or troglitazone) — Drug exposure will be inferred from prescription claims. Subjects who have been exposed to TZD for at least 6 months or at least 12 months will be considered for inclusion.
Drug: TZD + spironolactone — Subjects who have been exposed to TZD for at least 6 months or at least 12 months will be considered for inclusion.
  In order to be eligible for inclusion in this category, the prescription days supply for TZD and spirinolactone must overlap by at least 30 days.
Drug: TZD + amiloride — Subjects who have been exposed to TZD for at least 6 months or at least 12 months will be considered for inclusion.
  In order to be eligible for inclusion in this category, the prescription days supply for TZD and Amiloride must overlap by at least 30 days.

SUMMARY:
Treatment with thiazolidinediones (TZD) has recently been reported to possibly increase the risk of fractures in a randomized trial exploring the efficacy of rosiglitazone (RSG), metformin, or glyburide encompassing 4360 patients with type 2 diabetes.

It is hypothesized that spironolactone, a diuretic that is broadly used for the treatment of fluid retention and edema associated with TZD, has a potential protective effect against bone fractures. However, to our knowledge, this has not been tested in diabetic patients treated with TZD. Amiloride is another diuretic that shares with spironolactone the anti mineralocorticoid ion gated channels activity and will be analysed in this study with regard to possible protective effect against bone fracture in combination with TZD.

This study is a nested case-control study conducted among type 2 diabetes subjects exposed to TZD. The study aims to explore if the risk of fracture is reduced among type 2 diabetic subjects exposed to spironolactone and TZD. The study will compare the odds of any low impact fracture, and hand, foot, upper arm, wrist, and hip fracture incidence in subjects treated with TZD+spironolactone and TZD+amiloride compared to subjects treated with TZD only.

The study population will consist of type 2 diabetes patients aged 18 -65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one International Classification of Disease (ICD)-9 code for type 2 diabetes and have at least 6 months or at least 12 months of exposure to TZD (rosiglitazone [RSG], pioglitazone [PIO] or troglitazone) during their follow-up time available in the database.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* At least one ICD-9 code for type 2 diabetes
* At least 6 months or at least 12 months of exposure to TZD (RSG, PIO or troglitazone) during their follow-up time available in the database (The subject's study period begin date will be defined as the earliest date of their first TZD prescription. Subjects included in the study are required to have at least six months of follow-up time in the database prior to their first TZD prescription)

Exclusion Criteria:

* Subjects with a diagnosis of Paget's disease and osteomalacia
* A history of fracture, osteoporosis or cancer prior to the first prescription of TZD (study begin date)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of type 2 diabetes patients aged 18 -65 years old exposed to TZD for at least 6 months or at least 12 months. The study will use data from the US health claims database, the Ingenix Impact National Managed Care Database (Impact Database). The Impact Database system is a comprehensive, de-identified U.S. healthcare claims database that is representative of the non-elderly, insurance-carrying population. It includes 89.3 million lives from 1997 to 2008. Approximately 74 percent of all patients in the database have pharmacy benefits and, on average, 25 months of enrollment/claims information. The data are collected from over 46 different healthcare plans serving members across nine census regions.
Sampling Method: Non-Probability Sample
Enrollment: 98483 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- TZD 6-month Cohort (Including TZD 12-month Cohort): The study population consisted of type 2 diabetes patients 18-65 years old exposed to thiazolidinedione (TZD). To be eligible for the study, a subject must have had at least one International Classification of Disease (ICD)-9 code for type 2 diabetes and have at least 6 months of exposure to TZD (rosiglitazone [RSG], pioglitazone [PIO], or troglitazone) during their follow-up time available in the database. A subset of patients were followed for at least 12 months (Outcome measure results for this subset also presented). Dose information was not collected.
Period: Overall Study
Arm/Group | TZD 6-month Cohort (Including TZD 12-month Cohort)
Started | 98483
Completed | 98483
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TZD 6-month Cohort (Including TZD 12-month Cohort)
Number analyzed (Participants) | 98483
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37738
  Male | 60745

OUTCOME MEASURES:

1. Primary Outcome: Number of Low Impact Fractures in Males and Females After 6 Months of Exposure to TZD
Description: ICD-9 codes (805-807.4x, 808-810.xx, 812-829.xx) were captured from Uniform Billing-92 records and Health Care Finance Administration records. Case is defined as incident cases of fracture with an ICD-9 diagnostic code for any low impact fracture occurring after the study period begin date (earliest date of the first TZD prescription). For each subject defined as case, up to four controls were randomly selected from patients with type 2 diabetes exposed to TZD without a fracture diagnosis during follow-up and matched to cases on age (+ 5 years), gender, and year of fracture diagnosis.
Time Frame: From the earliest date of first TZD prescription to the fracture diagnosis date (Cases) or the end of follow-up in the database (Controls) between January 1, 1997 and December 31, 2008
Population: Type 2 diabetes patients 18-65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one ICD-9 code for type 2 diabetes and have at least 6 months of exposure to TZD (RSG, PIO, or troglitazone) during their follow-up time available in the database.
Measure: Number; unit: fractures
Groups:
- TZD Alone: Subjects with type 2 diabetes who had prescriptions for TZD only during their entire follow-up. Dose information was not collected.
- TZD+Spironolactone: Subjects with type 2 diabetes who had prescriptions for TZD and spironolactone during their entire follow-up. The prescription days supply for TZD and spirinolactone must overlap by at least 30 days. Dose information was not collected.
- TZD+Amiloride: Subjects with type 2 diabetes who had prescriptions for TZD and amiloride during their entire follow-up. The prescription days supply for TZD and amiloride must overlap by at least 30 days. Dose information was not collected.
- Other: Subjects with type 2 diabetes with exposure to TZD, but did not fit into the TZD Alone, TZD+Spironolactone, or TZD+Amiloride treatment groups during their entire follow-up. The prescription days supply for TZD and other drugs must overlap by at least 30 days. Dose information was not collected.
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 21621 | 397 | 43 | 3
fractures
  Case | 4325 | 105 | 12 | 1
  Control | 17296 | 292 | 31 | 2
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.13 to 1.78] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.93 to 1.52] — Adjusted Odds Ratio. Reference group TZD alone. Adjusted: age, liver disease, angina, renal and heart failure, asthma, stroke, epilepsy, RA, antihypertensives, statins, corticosteroids, antiepileptics, benzodiazepines, HRT, bisphosphonates
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.78 to 2.98] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.74 to 2.89] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.18 to 22.14] — Undadjusted Odds Ratio. Reference Group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.12 to 15.50] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Low Impact Fractures in Males and Females After 12 Months of Exposure to TZD
Description: as for outcome 1
Time Frame: From the earliest date of first TZD prescription to the fracture diagnosis date (Cases) or the end of follow-up in the database (Controls) between January 1, 1997 to December 31, 2008
Population: The study population consisted of type 2 diabetes patients aged 18 -65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one ICD-9 code for type 2 diabetes and have at least 12 months of exposure to TZD (RSG, PIO or troglitazone) during their follow-up time available in the database.
Measure: Number; unit: fractures
Groups:
- TZD Alone: Subjects with type 2 diabetes who had prescriptions for TZD during their entire follow-up. Dose information was not collected.
- TZD+Spironolactone: Subjects with type 2 diabetes who had prescriptions for TZD and spironolactone during their entire follow-up. The prescription days supply for TZD and amiloride must overlap by at least 30 days. Dose information was not collected.
- Other: Subjects with type 2 diabetes with exposure to TZD, but did not fit into any of the first 3 arms (TZD only, TZD+spironolacton, and TZD+amiloride) during their entire follow-up. The prescription days supply for TZD and other drugs must overlap by at least 30 days. Dose information was not collected.
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 13115 | 245 | 28 | 2
fractures
  Case | 2619 | 64 | 8 | 0
  Control | 10496 | 181 | 20 | 2
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.05 to 1.89] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.88 to 1.65] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.69 to 3.60] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.70 to 3.81] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Small numbers model didn't converge. Ref grp: TZD alone. Adjusted: age, liver disease, angina, renal and heart failure, asthma, stroke, epilepsy, RA, antihypertensives, statins, corticosteroids, antiepileptics, benzodiazepines, HRT, bisphosphonates

3. Secondary Outcome: Number of Fractures of the Hand, Foot, Upper Arm, and Wrist in Males and Females After 6 Months of Exposure to TZD
Description: ICD-9 codes (815.0x, 816.0x, 817.0x, 825.0x, 825.2x, 826.0x, 812.0x, 812.2x, 812.4x, 814.0x) were captured from UB-92 records and HCFA 1500 records. Case is defined as incident cases of fracture with an ICD-9 diagnostic code for hand, foot, upper arm, and wrist fracture after the study period begin date (earliest date of the first TZD prescription). For each case, up to four controls were randomly selected from patients with type 2 diabetes exposed to TZD without a fracture diagnosis during follow-up and matched on age (+ 5 yrs), gender, and year of fracture diagnosis.
Time Frame: as for outcome 2
Population: The study population consisted of type 2 diabetes patients aged 18 -65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one ICD-9 code for type 2 diabetes and have at least 6 months of exposure to TZD (RSG, PIO or troglitazone) during their follow-up time available in the database.
Measure: Number; unit: fractures
Groups:
- Other: Subjects with type 2 diabetes with exposure to TZD, but did not fit into any of the first 3 arms (TZD only, TZD+spironolactone, and TZD+amiloride) during their entire follow-up. The prescription days supply for TZD and other drugs must overlap by at least 30 days. Dose information was not collected.
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 10778 | 196 | 20 | 3
fractures
  Case | 2163 | 48 | 2 | 1
  Control | 8615 | 148 | 18 | 2
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.92 to 1.79] — Unadjusted Odds Ratio. Reference Group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.71 to 1.45] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.10 to 1.90] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.08 to 1.54] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.18 to 21.93] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.09 to 12.36] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Number of Fractures of the Hand, Foot, Upper Arm, and Wrist in Males and Females After 12 Months of Exposure to TZD
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: fractures
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 6400 | 123 | 12 | 2
fractures
  Case | 1285 | 29 | 0 | 0
  Control | 5115 | 94 | 12 | 2
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.80 to 1.88] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.62 to 1.57] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]

5. Secondary Outcome: Number of Hip Fractures Combined in Males and Females After 6 Months of Exposure to TZD
Description: ICD-9 codes (820.0x, 820.2x, 820.8x) were captured from UB-92 records and HCFA 1500 records. Case is defined as incident cases of fracture with an ICD-9 diagnostic code for hip fracture after the study period begin date (earliest date of the first TZD prescription). For each case, up to four controls were randomly selected from patients with type 2 diabetes exposed to TZD without a fracture diagnosis during follow-up and matched on age (+ 5 yrs), gender, and year of fracture diagnosis.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: fractures
Groups:
- Other: Subjects with type 2 diabetes with exposure to TZD, but did not fit into any of the first 3 arms (TZD only, TZD+spironolactone, and TZD+amiloride) during their entire follow-up. The prescription days supply for TZD and other drugs must overlap by at least 30 days
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 479 | 10 | 0 | 0
fractures
  Case | 92 | 6 |  |
  Control | 387 | 4 |  |
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 5.46, 95% CI 2-sided [1.53 to 19.45] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 3.19, 95% CI 2-sided [0.64 to 15.86] — Unadjusted Odds Ratio. Reference group TZD alone. Adjusted: age, liver disease, angina, renal and heart failure, asthma, stroke, epilepsy, RA, antihypertensives, statins, corticosteroids, antiepileptics, benzodiazepines, HRT, bisphosphonates
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]

6. Secondary Outcome: Number of Hip Fractures Combined in Males and Females After 12 Months of Exposure to TZD
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: fractures
Arm/Group | TZD Alone | TZD+Spironolactone | TZD+Amiloride | Other
Number analyzed (Participants) | 226 | 3 | 0 | 0
fractures
  Case | 44 | 2 |  |
  Control | 182 | 1 |  |
Statistical Analysis 1: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 7.26, 95% CI 2-sided [0.66 to 80.35] — Unadjusted Odds Ratio. Reference group: TZD alone
Statistical Analysis 2: Comparison: TZD Alone vs TZD+Spironolactone; Test type: Superiority or Other; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.03 to 96.47] — Adjusted Odds Ratio. Reference group: TZD alone. Adjusted: age, liver disease, angina, renal and heart failure, asthma, stroke, epilepsy, RA, antihypertensives, statins, corticosteroids, antiepileptics, benzodiazepines, HRT, bisphosponates
Statistical Analysis 3: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference Group: TZD alone
Statistical Analysis 4: Comparison: TZD Alone vs TZD+Amiloride; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 5: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Unadjusted Odds Ratio. Small numbers model didn't converge. Reference group: TZD alone
Statistical Analysis 6: Comparison: TZD Alone vs Other; Test type: Superiority or Other; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 2, analysis 6]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Groups:
- TZD 6-month Cohort: The study population consisted of type 2 diabetes patients 18-65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one ICD-9 code for type 2 diabetes and have at least 6 months of exposure to TZD (RSG, PIO, or troglitazone) during their follow-up time available in the database.
- TZD-12 Month Cohort: The study population consisted of type 2 diabetes patients 18-65 years old exposed to TZD. To be eligible for the study, a subject must have had at least one ICD-9 code for type 2 diabetes and have at least 12 months of exposure to TZD (RSG, PIO, or troglitazone) during their follow-up time available in the database.
Arm/Group | TZD 6-month Cohort | TZD-12 Month Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.